CLINICAL TRIAL: NCT06699251
Title: Effectiveness of Brief Intervention in Primary Care for Diverse Young People
Brief Title: Effectiveness of Brief Intervention in Primary Care for Diverse Young People (Chat)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: AltaMed Health Services Corporation (Other); University of Pittsburgh Medical Center (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-N0065
Record Dates: First submitted 2024-11-15; First posted 2024-11-21 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Adolescent Drinking; Cannabis Use
MeSH Terms: conditions — Underage Drinking | interventions — Choline O-Acetyltransferase

STUDY DESIGN:
Intervention Model Description: Enhanced Usual Care vs Chat Intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): When the online consent/assent form is completed, the teen will be sent a personalized link to complete their baseline survey. Upon survey completion, the teen will receive a link that has their electronic gift card payment, and the case manager will be notified that a particular ID has completed the survey. The case manager will be informed by study staff whether to schedule that ID for enhanced usual care (EUC) or the Chat intervention. If they are randomized as EUC, the informational brochure for the EUC will be handed to the teen during the visit or securely emailed to them. Whether the teen completes EUC or Chat, every teen will be followed by the RAND Survey Research Group to complete their paid follow-up web-based surveys based on timing of completion of their baseline survey.
  Interventions: Behavioral: Enhanced Usual Care
- Chat Intervention (Experimental): When the online consent/assent form is completed, the teen will be sent a personalized link to complete their baseline survey. Upon survey completion, the teen will receive a link that has their electronic gift card payment, and the case manager will be notified that a particular ID has completed the survey. The case manager will be informed by study staff whether to schedule that ID for enhanced usual care (EUC) or the Chat Intervention. If they are randomized as Chat Intervention, Chat will take place either via a virtual or in-person visit. Whether the teen completes EUC or Chat, every teen will be followed by the RAND Survey Research Group to complete their paid follow-up web-based surveys based on timing of completion of their baseline survey.
  Interventions: Behavioral: Chat

INTERVENTIONS:
Behavioral: Chat — Chat is a brief motivational interviewing intervention for partner clinic participants with an alcohol or cannabis use condition.
  Arms: Chat Intervention
Behavioral: Enhanced Usual Care — An informational brochure will be give to partner clinic participants with an alcohol or cannabis use condition.
  Arms: Enhanced Usual Care

SUMMARY:
Brief motivational interviewing intervention to address alcohol use among diverse teens 12-17.

DETAILED DESCRIPTION:
The six-item CRAFFT will be used to screen teens at our partner clinics for risky AC use. For those that screen in as at-risk and express interest in the study, the teen's case manager will complete an online consent/assent form with the parent and teen that contains contact information for the teen so that investigators can follow up with the teen for surveys and intervention delivery or for providing an informational brochure. When the online consent/assent form is completed, the teen will be sent a personalized link to complete their baseline survey. Upon survey completion, the teen will receive a link that has their electronic gift card payment, and the case manager will be notified that a particular ID has completed the survey. The case manager will be informed by study staff whether to schedule that ID for enhanced usual care (EUC) or the Chat intervention. Investigators expect each teen to be scheduled within 30 days of completing their baseline survey to receive EUC or Chat. The informational brochure for the EUC will be handed to the teen during the visit or securely emailed, and Chat could take place either via a virtual or in-person visit. Whether or not the teen completes EUC or Chat, every teen will be followed by the RAND Survey Research Group to complete their follow-up web-based surveys based on timing of completion of their baseline survey. Teens will receive gift card incentives for completing the 3-month, 6-month, and 12-month surveys. Investigators will begin recruitment in month 9 of the project. Briefly, investigators expect to recruit from study month 9 to month 42 for the baseline survey. Investigators expect the Chat intervention to occur from months 9 to 42 the 3-month follow-up from months 12 to 45, 6-month from months 15 to 48, and the 12-month from months 21 to 53. Out of an anticipated 5,644 clients that our partner clinics will screen, investigators expect approximately 847 (15%) to screen in as at-risk on the CRAFFT and anticipate that approximately 500 (~60%) will consent into the study.

ELIGIBILITY:
Inclusion Criteria:

* receive health care at one of two participating health systems
* aged 12-17
* screen positive for being at risk for alcohol or cannabis use using the CRAFFT

Exclusion Criteria:

* if they don't meet the inclusion criteria, they will be excluded

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-07-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Alcohol - change in frequency of use | Baseline to 3 months
  We will assess both the number of times participants have used alcohol in the past three months (from none to 31 or more times) and the number of days in the past month participants report use of alcohol.
Alcohol - change in frequency of use | 3 months to 6 months
  We will assess both the number of times participants have used alcohol in the past three months (from none to 31 or more times) and the number of days in the past month participants report use of alcohol.
Alcohol - change in frequency of use | 6 months to 12 months
  We will assess both the number of times participants have used alcohol in the past six months (from none to 31 or more times) and the number of days in the past month participants report use of alcohol.
Cannabis - change in frequency of use | Baseline to 3 months
  We will assess both the number of times participants have used cannabis in the past three months (from none to 31 or more times) and the number of days in the past month participants report use of cannabis.
Cannabis - change in frequency of use | 3 months to 6 months
  We will assess both the number of times participants have used cannabis in the past three months (from none to 31 or more times) and the number of days in the past month participants report use of cannabis.
Cannabis - change in frequency of use | 6 months to 12 months
  We will assess both the number of times participants have used cannabis in the past six months (from none to 31 or more times) and the number of days in the past month participants report use of cannabis.
Alcohol - change in consequences of use | Baseline to 3 months
  Alcohol consequences (e.g., blacking out, regretted sexual situation) will be assessed with the Brief Young Adult Alcohol Consequences Questionnaire (0 to 20 or more times, with higher scores indicating a worse outcome).
Alcohol - change in consequences of use | 3 months to 6 months
  Alcohol consequences (e.g., blacking out, regretted sexual situation) will be assessed with the Brief Young Adult Alcohol Consequences Questionnaire (0 to 20 or more times, with higher scores indicating a worse outcome).
Alcohol - change in consequences of use | 6 months to 12 months
  Alcohol consequences (e.g., blacking out, regretted sexual situation) will be assessed with the Brief Young Adult Alcohol Consequences Questionnaire (0 to 20 or more times, with higher scores indicating a worse outcome).
Cannabis - change in consequences of use | Baseline to 3 months
  Cannabis consequences (e.g., poor memory, too much time using) will be assessed with the Brief Marijuana Consequences Questionnaire (0 to 20 or more times, with higher scores indicating a worse outcome).
Cannabis - change in consequences of use | 3 months to 6 months
  Cannabis consequences (e.g., poor memory, too much time using) will be assessed with the Brief Marijuana Consequences Questionnaire (0 to 20 or more times, with higher scores indicating a worse outcome).
Cannabis - change in consequences of use | 6 months to 12 months
  Cannabis consequences (e.g., poor memory, too much time using) will be assessed with the Brief Marijuana Consequences Questionnaire (0 to 20 or more times, with higher scores indicating a worse outcome).

SECONDARY OUTCOMES:
Alcohol - change in time spent around peers | Baseline to 3 months
  Participants will be asked how often they are with people their age who are using alcohol (1=never to 4=often).
Alcohol - change in time spent around peers | 3 months to 6 months
  Participants will be asked how often they are with people their age who are using alcohol (1=never to 4=often).
Alcohol - change in time spent around peers | 6 months to 12 months
  Participants will be asked how often they are with people their age who are using alcohol (1=never to 4=often).
Cannabis - change in time spent around peers | Baseline to 3 months
  Participants will be asked how often they are with people their age who are using cannabis (1=never to 4=often).
Cannabis - change in time spent around peers | 3 months to 6 months
  Participants will be asked how often they are with people their age who are using cannabis (1=never to 4=often).
Cannabis - change in time spent around peers | 6 months to 12 months
  Participants will be asked how often they are with people their age who are using cannabis (1=never to 4=often).
Alcohol - change in motivation to change use | Baseline to 3 months
  We will measure motivation to change use by asking participants where they may be in their thinking about reducing or quitting their alcohol use using a scale of 1-10 where 1 = "I have quit using alcohol and will never go back" and 10 = "I enjoy using alcohol and have decided never to change it."
Alcohol - change in motivation to change use | 3 months to 6 months
  We will measure motivation to change use by asking participants where they may be in their thinking about reducing or quitting their alcohol use using a scale of 1-10 where 1 = "I have quit using alcohol and will never go back" and 10 = "I enjoy using alcohol and have decided never to change it."
Alcohol - change in motivation to change use | 6 months to 12 months
  We will measure motivation to change use by asking participants where they may be in their thinking about reducing or quitting their alcohol use using a scale of 1-10 where 1 = "I have quit using alcohol and will never go back" and 10 = "I enjoy using alcohol and have decided never to change it."
Cannabis - change in motivation to change use | Baseline to 3 months
  We will measure motivation to change use by asking participants where they may be in their thinking about reducing or quitting their cannabis use using a scale of 1-10 where 1 = "I have quit using cannabis and will never go back" and 10 = "I enjoy using cannabis and have decided never to change it."
Cannabis - change in motivation to change use | 3 months to 6 months
  We will measure motivation to change use by asking participants where they may be in their thinking about reducing or quitting their cannabis use using a scale of 1-10 where 1 = "I have quit using cannabis and will never go back" and 10 = "I enjoy using cannabis and have decided never to change it."
Cannabis - change in motivation to change use | 6 months to 12 months
  We will measure motivation to change use by asking participants where they may be in their thinking about reducing or quitting their cannabis use using a scale of 1-10 where 1 = "I have quit using cannabis and will never go back" and 10 = "I enjoy using cannabis and have decided never to change it."
Change in use of behavioral health care services | Baseline to 3 months
  We will measure use of behavioral health care services (separate items for mental health and substance use), including whether there are unmet needs for behavioral health services (i.e., perceived a need to get treatment but didn't get it) and perceived reasons for those unmet needs (e.g., stigma, transportation, cost).
Change in use of behavioral health care services | 3 months to 6 months
  We will measure use of behavioral health care services (separate items for mental health and substance use), including whether there are unmet needs for behavioral health services (i.e., perceived a need to get treatment but didn't get it) and perceived reasons for those unmet needs (e.g., stigma, transportation, cost).
Change in use of behavioral health care services | 6 months to 12 months
  We will measure use of behavioral health care services (separate items for mental health and substance use), including whether there are unmet needs for behavioral health services (i.e., perceived a need to get treatment but didn't get it) and perceived reasons for those unmet needs (e.g., stigma, transportation, cost).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. D'Amico, PhD, Principal Investigator — RAND; Alina I Palimaru, PhD, Principal Investigator — RAND
Locations (2):
- United States (2):
  - AltaMed Health Services, Commerce, California
  - University of Pittsburgh Medical Center Children's Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT06699251/Prot_SAP_000.pdf